CLINICAL TRIAL: NCT00526188
Title: A Multicenter, Open-label Phase III Study of the Efficacy and Safety of Primovist as a Contrast Agent for Enhanced MR Imaging of Focal Liver Lesions in Chinese Patients
Brief Title: Efficacy and Safety of Primovist in Chinese Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 91531; 310682 (Other: Company internal)
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Results first posted 2009-12-30 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Known or Suspected Focal Liver Lesions
Keywords: Primovist; Chinese patients; Liver MRI
MeSH Terms: interventions — gadolinium ethoxybenzyl DTPA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gadoxetic Acid Disodium (Primovist, BAY86-4873) (Experimental): Bolus injection of 0.025 mmol/kg body weight (0.1 ml/kg BW) of Gadoxetic Acid Disodium (Primovist, BAY86-4873). Single i.v. injection during MRI procedure, with one contrast-enhanced MRI procedure per patient
  Interventions: Drug: Gadoxetic Acid Disodium (Primovist, BAY86-4873)

INTERVENTIONS:
Drug: Gadoxetic Acid Disodium (Primovist, BAY86-4873) — Bolus injection of 0.025 mmol/kg body weight (0.1 ml/kg BW) of Gadoxetic Acid Disodium (Primovist, BAY86-4873). Single i.v. injection during MRI procedure, with one contrast-enhanced MRI procedure per patient

SUMMARY:
Participants who had been diagnosed or suspected by doctors to have focal liver lesions that need further evaluation in order to make an accurate diagnosis. Participants would need to have an enhanced magnetic resonance imaging (MRI) scan so that doctors could have further information about the number and characteristics of the focal liver lesions.

Participants were invited to take part in this clinical study. The purpose of this study was to evaluate Primovist, which is a liver-specific MRI contrast medium, on the efficacy of lesion detection and characterization, and tolerability in Chinese patients with known or suspected focal liver lesions.

Primovist, the investigational drug in this study, is a liver-specific MRI contrast medium developed by Bayer Schering Pharma AG. Its active substance is Gd-EOB-DTPA. Primovist was first approved in 2004 in Sweden followed by an approval in the European community, in Switzerland and Australia in the same year.

Procedures:

Before entry into the study and after entry of the study a physical examination was conducted, blood pressure and heart rate were measured, blood and urine samples were taken. Current medications and medical conditions (including suspected pregnancy) and medical and surgical history were elicited by doctors.

After entry into the study, participants were scheduled to have an MRI examination, which lasted about 25-35 minutes.

During the MRI examination, an initial MRI scan without contrast was acquired which followed by another MRI series after the intravenous administration of Primovist.

The following day participants were asked to return to the hospital for a follow-up safety evaluation.

Possible Benefit Participants were scheduled to receive an enhanced magnetic resonance imaging scan. Clinical studies indicated that Primovist increased the efficacy of detection and characterization of focal liver lesions by providing better contrast between the focal liver lesions and surrounding normal tissue. Primovist were shown to provide additional information regarding existence, number and characterization (lesion or non-lesion, malignant or benign) of these abnormalities.

Based on the experience with patients given Primovist, some adverse reactions were observed.

Most of undesirable effects were transient and of mild to moderate intensity. The most commonly noted adverse events (AEs) in subjects receiving Primovist for MRI were nausea and headache with an incidence of 1.1%. Other AEs that occurred in 0.5% of the subject population were feeling hot (0.8%), back pain (0.6%) and dizziness (0.5%).

All other AEs occurred in less than 0.5% of the patients, e.g. anxiety; coughing; eye disorder; fever; flatulence; generalized spasm; hypertension; injection site symptoms including edema, inflammation, and reaction; lightheadedness; parosmia; postural hypotension; taste perversion, motoric unrest; acute respiratory distress; fatigue; malaise; vomiting; palpitations, erythema, chest pain and back pain.

Coldness, warmth or pain at the injection site, injection site reaction, and injection site accumulation of fluid were rare. In very rare cases strong allergy-like reactions ranging to shock may occur.

Post-marketing tachycardia and restlessness have been reported. As in the case of other investigational drugs, there may also be unforeseen side effects.

Additional information concerning all Gadolinium- based contrast agents Primovist contains the rare earth metal gadolinium as active ingredient. There have been reports of nephrogenic systemic fibrosis (NSF) associated with use of some gadolinium-containing contrast agents (especially Omniscan) in patients with severe renal impairment. NSF is a systemic disease characterised by formation of connective tissue in the skin, which becomes thickened and hard, sometimes leading to contractures and joint immobility. The clinical course is usually progressive and currently no treatment is available. To date NSF has only been reported in association with some Gd-containing contrast agents, but the role of these contrast agents in the overall pathogenesis of the disease is still not completely understood.

No reports of patients with NSF after administration of Primovist® are known. The risk to trigger NSF in risk patients with severe renal impairment is considered to be low for Primovist® due to the low dose given and the additional excretion via feces. Furthermore the participation of patients with severe renal impairment are excluded from this study.

In case the participants were suffering from renal insufficiency, they were told to tell their doctors prior to application of the contrast agent. In case the participants experienced any new alterations of the skin following the administration of the contrast agent, they were told to contact their doctors as soon as possible after they had recognized these symptoms.

DETAILED DESCRIPTION:
Adult Chinese patients with known focal or suspected liver lesions, referred for magnetic resonance imaging (MRI) for further diagnostic work-up, who have undergone or are scheduled to undergo a defined SOR procedure, within one month before or after the study MRI.

The data for the Secondary Outcome Measure "Lesion size and location" has been documented but not analyzed. The data for the Secondary Outcome Measure "Safety" are reflected in the Adverse Event section.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 75 years of age inclusive.
* Patients (men or women) with at least one focal liver lesion, either identified or suspected by ultrasound (US), Computed Tomography (CT)/spiral-CT, conventional angiography, CT-angiography (CTA), CT-arterioportography (CTAP) or unenhanced / contrast-enhanced MRI* within 2 months before entering the study

For reference, the following pathologies will meet the definition of 'focal liver lesions':

* Hepatocellular carcinoma
* Cholangiole carcinoma
* Metastasis
* Focal lymphoma
* Adenoma
* Focal nodular hyperplasia
* Hemangioma
* Abscess
* Focal liver fibrosis
* Regenerative nodules
* Focal fatty infiltration
* Hydatid cyst
* Liver cyst
* Focal sparing in fatty liver
* Others
* Patients willing to undergo study procedures including safety follow-up
* Patients who have undergone or who are scheduled to undergo the defined procedure for SOR within one month before or after the study MRI
* Women of child-bearing potential with negative urine pregnancy test result within 24 hours before contrast medium (CM) injection
* Patients who are fully informed about the study and have signed the informed consent form

Exclusion Criteria:

* Patients who have previously entered this study
* Patients who have received any contrast material within 24 hours before injection with study drug, or who are scheduled to receive any contrast material within 24 hours after injection
* Patients who are, or suspected to be, nursing
* Patients who require emergency treatment
* Patients with severely impaired hepatic or renal functions (e.g. serum glutamic-pyruvic transaminase (SGPT) twice the upper limit of reference range, acute renal failure)
* Patients who are clinically unstable and whose clinical course during the observation period is unpredictable (e.g. due to previous surgery, acute myocardial infarction)
* Patients with any physical or mental status that interferes with the signing of informed consent
* Patients with known anaphylactoid or anaphylactic reaction to any contrast media or hypersensitivity to any allergen including drugs
* Patients with a contraindication for MRI
* Patients who are scheduled for liver biopsy/surgery or other surgeries within 24 hours after injection with contrast media, or who would have a biopsy within 24 hours before planned injection with contrast media
* Patients who are likely to have any therapy or change in therapy between the study MRI and the procedures for the SOR

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2007-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (5):
- China (5):
  - Nanjing, Jiangsu
  - Suzhou, Jiangsu
  - Xi'an, Shaanxi
  - Beijing
  - Shanghai

REFERENCES:
- [Result] Zeng MS, Ye HY, Guo L, Peng WJ, Lu JP, Teng GJ, Huan Y, Li P, Xu JR, Liang CH, Breuer J. Gd-EOB-DTPA-enhanced magnetic resonance imaging for focal liver lesions in Chinese patients: a multicenter, open-label, phase III study. Hepatobiliary Pancreat Dis Int. 2013 Dec;12(6):607-16. doi: 10.1016/s1499-3872(13)60096-x. PMID 24322746

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was 20 Aug 2007 to 30 Aug 2008.
Pre-assignment Details: 247 Chinese patients were recruited and screened. Among these, 13 patients were screening failures: withdrawal of consent (7 patients), non-fulfillment of the inclusion and exclusion criteria (3 patients), other reasons (3 patients). The remaining 234 patients received the study drug and were included in the safety analysis set.
Period: Overall Study
Arm/Group | Gadoxetic Acid Disodium (Primovist, BAY86-4873)
Started | 234
Completed | 234
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gadoxetic Acid Disodium (Primovist, BAY86-4873)
Number analyzed (Participants) | 234
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (11.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79
  Male | 155
Characterization of first liver lesion type of referral diagnosis [Number; unit: participants]
  Hepatocellular carcinoma | 47
  Cholangiocarcinoma | 1
  Metastasis | 58
  Focal nodular hyperplasia | 14
  Hemangioma | 42
  Abscess | 2
  Focal fatty infiltration | 1
  Liver cyst | 13
  Inflammation | 1
  Harmatoma | 1
  Infection | 1
  Inflammatory pseudotumor | 2
  Not assessable | 51
Characterization of second liver lesion type of referral diagnosis [Number; unit: participants]
  No second liver lesion type | 191
  Hepatocellular carcinoma | 3
  Metastasis | 5
  Hemangioma | 7
  Hydatid cyst | 1
  Liver cyst | 23
  Calcification | 1
  Inflammatory pseudotumor | 1
  Not assessable | 2
Characterization of third liver lesion type of referral diagnosis [Number; unit: participants]
  No third liver lesion type | 231
  Hemangioma | 1
  Liver cyst | 1
  Calcification | 1

OUTCOME MEASURES:

1. Primary Outcome: Difference in Sensitivity of Lesion Detection in MRI Images (Post-contrast MRI Minus Pre-contrast MRI) Measured as Percentage Points
Description: Three Blinded Readers performed lesion detection in pre- and post-contrast MRI image sets. Per Blinded Reader/image set combination, sensitivity of lesion detection was calculated, as: (number of lesions detected in the reader/image set combination)/(number of lesions in Standard of Reference)*100%. Then, difference in sensitivity of lesion detection for post- minus pre-contrast MRI images (in percentage points) was calculated for each Blinded Reader.
Time Frame: Post administration assessment of study images (i.e. on the same day of treatment by the investigators and at the end of patient enrollment of the study from 29 September to 18 November 2008 by the Blinded Readers).
Population: All participants from the per protocol set with pre- and post-contrast MRI image sets evaluable for all blinded readers, with at least 1 lesion in the Standard of Reference (SOR)
Measure: Mean (95% Confidence Interval); unit: Percentage points
Arm/Group | Gadoxetic Acid Disodium (Primovist, BAY86-4873)
Number analyzed (Participants) | 176
Percentage points
  BR 1: Dif. in sens. post- minus pre-contrast MRI | 8.65 [4.82 to 12.47]
  BR 2: Dif. in sens. post- minus pre-contrast MRI | 12.23 [7.60 to 16.87]
  BR 3: Dif. in sens. post- minus pre-contrast MRI | 7.50 [2.84 to 12.17]
Statistical Analysis 1: Comparison: Gadoxetic Acid Disodium (Primovist, BAY86-4873); Difference in sensitivity of lesion detection between post- and pre-contrast MRI image set was calculated. Null hypothesis: No difference between post- and pre-contrast MRI image set. Test was performed based on a normal-approximated confidence interval (CI) for the average blinded reader difference. This CI had a confidence level of 95% and was two-sided. The study was planned with a power of 80%; Test type: Superiority or Other; Test performed based on the 95% CI; Mean Difference (Final Values) = 9.46, 95% CI [6.00 to 12.93] — Comparison was post-contrast MRI minus pre-contrast MRI

2. Secondary Outcome: Difference in Sensitivity of Lesion Detection in MRI Images (Post-contrast MRI Minus Pre-contrast MRI) Assessed by Investigators Measured in Percentage Points
Description: The on-site investigators performed lesion detection in pre- and post-contrast MRI image sets. Per image set, sensitivity of lesion detection was calculated, as: (number of lesions detected in image set)/(number of lesions in Standard of Reference)*100%. Then, difference in sensitivity of lesion detection for post- minus pre-contrast MRI (in percentage points) was calculated.
Time Frame: as for outcome 1
Population: All participants from the per protocol set, with at least 1 lesion in the Standard of Reference (SOR).
Measure: Mean (95% Confidence Interval); unit: Percentage points
Arm/Group | Gadoxetic Acid Disodium (Primovist, BAY86-4873)
Number analyzed (Participants) | 177
Percentage points | 4.81 [1.84 to 7.78]
Statistical Analysis 1: Comparison: Gadoxetic Acid Disodium (Primovist, BAY86-4873); Difference in sensitivity of lesion detection between post- and pre-contrast MRI image sets, based on investigators assessments was calculated. Null hypothesis: No difference between post and pre contrast MRI image set. Test was performed based on a normal-approximated confidence interval (CI) for the investigators difference. This CI had a confidence level of 95% and was two-sided; Test type: Superiority or Other; Test performed based on the 95% CI; Mean Difference (Final Values) = 4.81, 95% CI [1.84 to 7.78] — Comparison was post-contrast MRI minus pre-contrast MRI (for investigator's result)

3. Secondary Outcome: Difference in Precision of Lesion Characterization (Combined Pre- and Post-contrast Minus Pre-contrast MRI) Measured in Percentage Points
Description: Three Blinded Reader performed lesion characterization in pre- and combined pre-/post-contrast MRI image set. Per Blinded Reader/image set combination, precision of lesion characterization was calculated: (number of unique Standard of Reference-matched characterizations detected for the Reader/image set combination)/(number of unique lesion characterizations in Standard of Reference)*100%. Then, difference in precision of lesion characterization for post- minus combined pre-/post-contrast MRI (in percentage points) was calculated for each Blinded Reader.
Time Frame: as for outcome 1
Population: All participants from the per protocol set with pre- and combined pre- and post- contrast MRI image sets evaluable for all blinded readers, with at least 1 lesion characterization in the Standard of reference (SOR)
Measure: Mean (95% Confidence Interval); unit: Percentage points
Arm/Group | Gadoxetic Acid Disodium (Primovist, BAY86-4873)
Number analyzed (Participants) | 165
Percentage points
  BR1: Dif. in prec. pre-/post- minus pre-contrast | 13.64 [7.80 to 19.47]
  BR2: Dif. in prec. pre-/post- minus pre-contrast | 9.55 [3.13 to 15.96]
  BR3: Dif. in prec. pre-/post- minus pre-contrast | 10.91 [5.32 to 16.50]
Statistical Analysis 1: Comparison: Gadoxetic Acid Disodium (Primovist, BAY86-4873); Difference in precision of lesion characterization between combined pre and post contrast MRI and pre contrast MRI image set was calculated. Null hypothesis: No difference between combined pre- and post-contrast MRI and pre contrast MRI image set. Test was performed based on a normal-approximated confidence interval (CI) for the average blinded reader difference. This CI had a confidence level of 95% and was two-sided; Test type: Superiority or Other; Test performed based on the 95% CI; Mean Difference (Final Values) = 11.36, 95% CI [7.45 to 15.28] — Comparison was combined pre- and post-contrast MRI minus pre-contrast MRI

ADVERSE EVENTS:
Arm/Group | Gadoxetic Acid Disodium (Primovist, BAY86-4873)
Serious Adverse Events (participants affected / at risk) | 0/234
Other Adverse Events (participants affected / at risk) | 20/234
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gadoxetic Acid Disodium (Primovist, BAY86-4873) (N=234)
Blood pressure systolic increased (Investigations) | 1
Hypertension (Vascular disorders) | 4
Blood pressure diastolic increased (Investigations) | 1
Hypotension (Vascular disorders) | 2
Blood lactate dehydrogenase increased (Investigations) | 3
Blood glucose increased (Investigations) | 2
Injection site pain (General disorders) | 1
Nausea (Gastrointestinal disorders) | 2
White blood cell count decreased (Investigations) | 2
Blood bilirubin increased (Investigations) | 3
Blood phosphorus increased (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less